CLINICAL TRIAL: NCT01232400
Title: Adrenergic Blockade After Subarachnoid Hemorrhage
Brief Title: Study to Evaluate Esmolol (Brevibloc) to Manage Cardiac Function in Patients With Subarachnoid Hemorrhage
Acronym: ABASH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn. Design not feasible.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, William J Meurer, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM31297
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Subarachnoid Hemorrhage
Keywords: subarachnoid hemorrhage; esmolol; cardiac function; cardiac electrophysiology
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- esmolol (Experimental): Esmolol will be used preferentially to control hypertension.
  Interventions: Drug: Esmolol
- Standard care (No Intervention): Standard care for SAH includes other hypertensives such as nicardipine.

INTERVENTIONS:
Drug: Esmolol — The initial esmolol infusion will be 50 mcg/kg/minute IV. This will be increased by 25 mcg/kg/minute every 15 minutes until one of the following situations is reached:
  1. Heart rate less than 70 bpm.
  2. Systolic blood pressure less than 120 mmHg
  3. Maximum dose of esmolol of 200 mcg/kg/minute is reached.
  Other Names: Brevibloc
  Arms: esmolol

SUMMARY:
The purpose of this study is to evaluate the clinical effect of esmolol treatment on cardiac function and electrophysiology; to assess the effects of esmolol treatment on serum adrenergic and cardiac biomarkers; to explore the safety of esmolol treatment shortly after subarachnoid hemorrhage (SAH). Patients will be followed for a maximum of 1 month after the index SAH. The primary outcome will be change in systolic function - ejection fraction by Simpson's rule (baseline versus Day 7 +/- 2 after SAH).

DETAILED DESCRIPTION:
Subarachnoid hemorrhage (SAH) remains one of the most devastating forms of stroke. Over 25% of all stroke related potential years of life lost are from SAH. Outcomes are adversely affected by secondary ischemia from cerebral vasospasm, along with cardiac complications. Trials performed in patients with SAH have demonstrated benefit after the administration of beta blockers - reducing mortality nearly in half; but concerns over diminishing cerebral perfusion inhibited the widespread adoption of this therapy. Our specific aims are as follows: 1. To evaluate the clinical effect of esmolol treatment on cardiac systolic and diastolic function, along with cardiac electrophysiology; 2. To assess the effects of esmolol treatment on serum adrenergic and cardiac biomarkers; 3. To explore the safety of esmolol shortly after SAH. The primary outcome will be change in systolic function - ejection fraction by Simpson's rule (baseline versus Day 7 +/- 2 after SAH).

ELIGIBILITY:
Inclusion Criteria:

* Subarachnoid hemorrhage presumed to be the result of ruptured aneurysm
* Age 18 years old or greater
* Able to enroll within 24 hours of onset of symptoms
* Systolic blood pressure over 140 mm Hg OR administration of antihypertensives after presentation

Exclusion Criteria:

* Withdrawal of life support imminent (within six hours)
* Known heart failure or cardiomyopathy AND ejection fraction 35% or below
* Prisoner or pregnant female
* Ongoing vasopressor administration to maintain SBP, or clinical suspicion of left ventricular failure
* Clinically important arrhythmias (history of cardiac arrest or ventricular arrhythmias), conduction abnormalities (Mobitz Type 2, 3rd degree AV block, or symptomatic Mobitz 1 without pacemaker), clinical cardiogenic shock, or overt clinical heart failure
* Active bronchospastic disease (ongoing bronchospasm after SAH presentation or current treatment with oral corticosteroids for asthma or obstructive lung disease)
* End stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change in high sensitivity troponin | Peak to nadir within 7 days

SECONDARY OUTCOMES:
Mean difference in time weighted average amount of cerebral perfusion pressure below 60 mmHg. | Measured for 4 days from index SAH
Proportion experiencing serious adverse event: hypotension requiring vasopressor (excluding during anesthesia), neurological deterioration, serious bronchospasm, and in hospital case fatality. | Measured during index hospitalization or first 30 days from index SAH
Disability (30 days +/-7). | 30 days from index SAH
Change in serum norepinephrine level from peak to nadir | Baseline versus 4th day after index SAH
Change in corrected QT interval | First week after presentation for index SAH
Proportion with echocardiographic wall motion abnormalities at baseline and day 7 +- 2 | First week after presentation.
Proportion with electrocardiographic abnormalities cumulative through day 7 | Baseline, and at first week after presentation.
Proportion with depressed ejection fraction on initial echocardiogram 36 - 49% | Baseline (within 24 hours of presentation for index SAH)
Proportion with life-threatening arrhythmias or cardiac arrest | Measured through end of index hospitalization (approximately 30 days maximum)
Change in serum troponin and BNP levels from peak to nadir | baseline through end of hospitalization
Proportion with abnormal 30-day echocardiogram | 30 days post index SAH
Proportion with symptomatic cerebral vasospasm | baseline until end of hospitalization
Proportion with radiographic cerebral vasospasm | baseline until end of hospitalization
Change in systolic function - ejection fraction by Simpson's rule (baseline vs Day 7 +/- 2) | 5-7 days

CONTACTS AND LOCATIONS:
Overall Officials: William J Meurer, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States